CLINICAL TRIAL: NCT03854617
Title: A Randomized, Open-label, Parallel Study to Evaluate the Efficacy and Safety of Oral Navelbine in Female Patients With HER2-Negative Metastatic Breast Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of Oral Navelbine in Female Patients With HER2-Negative Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Binghe Xu, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC2
Record Dates: First submitted 2019-02-19; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Human Epidermal Growth Factor 2 Negative Carcinoma of Breast
Keywords: oral Navelbine; Metastasis Breast Cancer; metronomic chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral NVB Metronomic (Experimental): 50mg three times weekly on Mondays (or Tuesdays), Wednesdays (or Thursdays) and Friday (or Saturdays). A cycle is a 3 weeks period.
  Interventions: Drug: Oral NVB Metronomic
- Oral NVB Weekly (Active Comparator): 60mg/m2 weekly for cycle 1 and 80mg/m2 weekly for subsequent cycles in the absence of grade 3 or 4 toxicity. A cycle is a 3 weeks period.
  Interventions: Drug: Oral NVB Weekly

INTERVENTIONS:
Drug: Oral NVB Metronomic — 50mg three times weekly on Mondays (or Tuesdays), Wednesdays (or Thursdays) and Friday (or Saturdays). A cycle is a 3 weeks period.
  Other Names: Oral Navelbine Metronomic
  Arms: Oral NVB Metronomic
Drug: Oral NVB Weekly — 60mg/m2 weekly for cycle 1 and 80mg/m2 weekly for subsequent cycles in the absence of grade 3 or 4 toxicity. A cycle is a 3 weeks period
  Other Names: Oral Navelbine Weekly
  Arms: Oral NVB Weekly

SUMMARY:
This is a randomized, open-label, parallel, multi-center study, aims to evaluate the efficacy and safety of metronomic chemotherapy with oral Navelbine versus intermittent oral Navelbine in female patients with HER2 negative Metastasis Breast Cancer.

DETAILED DESCRIPTION:
1. The significant efficacy and good safety profile of Vinorelbine in the treatment of advanced breast cancer are accepted.
2. Oral NVB presents absolute bioavailability of 40% and oral availability allows to use different schedules and the endothelial cell functionality and motility are interfered at very low drug concentration
3. Oral NVB at 50 mg three times a week (Monday-Wednesday-Friday) has been tested in phase Ia/Ib/II trials, highlighting the excellent safety of this scheme combined with an interesting activity in various European countries.
4. The study aims to evaluate the efficacy and safety of metronomic chemotherapy with oral Navelbine versus intermittent oral Navelbine in female patients with HER2 negative Metastasis Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with life expectancy ≥ 3 months, age ≥ 18 years at the time informed consent is signed.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 as assessed within 21 days prior to randomization (Appendix ).
* Subjects with HER2 negative metastasis breast cancer, source documented, defined as per American Society of Clinical Oncology - College of American Pathologists (ASCO/CAP) guidelines (Appendix ).
* Subjects with measurable metastatic disease defined by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) guidelines (Appendix ) .
* Subjects may previously exposed to anthracyclines (e.g. doxorubicin, epirubicin) and/or taxanes (e.g., paclitaxel, docetaxel) including:

  * Subject has been pretreated in the adjuvant or neoadjuvant setting with anthracyclines and/or taxanes before breast cancer relapsing;
  * Subjects has experienced treatment failure while receiving or after completing anthracycline- and/or taxane- based chemotherapy;
  * Subjects who are not suitable for the choice of anthracycline- and/or taxane- based chemotherapy as first-line treatment in the judgment of investigator.
* Prior radiotherapy must have completed before randomization, with full recovery from acute radiation side effects. An interval of less than 4 weeks after radiotherapy was not allowed.Concurrent limited field radiation therapy (RT) is allowed. At least one measurable lesion must be completely outside the radiation portal in accordance with RECIST 1.1 guidelines;
* At least 30 days from major surgery before randomization, with full recovery;
* Adequate bone marrow function as evidenced by the following:

  * Absolute Neutrophil Count (ANC) ≥ 1500/mm2;
  * Platelets ≥ 100,000/mm2;
  * Hemoglobin (Hb) ≥ 10 g/dL.
* Adequate liver function as evidenced by the following:

  * Total serum bilirubin ≤ 1.5 times upper limit of normal range (ULN);
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 times ULN (if hepatic metastases present ≤ 5.0 times ULN);
  * Alkaline phosphatase < 5 x ULN.
* Adequate renal function as evidenced by the following:

  -Creatinine clearance > 40 mL/min (by Cockcroft-Gault).
* Women of child-bearing potential must have a negative pregnancy test (urine or serum) within 7 days of randomization and agree to take an adequate contraceptive measure.
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
* Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* History of, or current active cancer other than breast cancer, with the exception of curatively resected non-melanomatous skin cancer, curatively treated cervical carcinoma in situ, or other primary solid tumors curatively treated with no known active disease present and no curative treatment administered for the last 3 years.
* Patients with medical conditions that the only manifestation is hydrothorax, ascites, bone lesions or other un-measurable diseases.
* Subjects with visceral crisis in the judgment of investigator. Visceral crisis is defined as severe organ dysfunction as assessed by signs and symptoms, laboratory studies, and rapid progression of disease. Visceral crisis is not the mere presence of disease of visceral metastases, but implies important visceral compromise leading to a clinical indication for a more rapidly efficacious therapy, particularly since chemotherapy option at progression will probably not be possible.
* Malabsorption syndrome or disease significantly affecting gastro-intestinal function or major resection of the stomach or proximal small bowel that could affect absorption of Oral NVB.
* Subjects with dysphagia, or inability to swallow the tablets.
* Subjects with symptoms suggesting central nervous system (CNS) involvement or leptomeningeal metastases, any suspicious sins or symptoms of CNS involvement or leptomeningeal metastases should be excluded by CT or MRI scans.
* Other serious illness or medical conditions by the investigator during screening:

  * Clinically significant cardiac disease;
  * Unstable diabetes;
  * Uncontrolled hypercalcemia;
  * Clinically significant active infections (current or in the last two weeks).
* Previous organ allograft.
* Current peripheral neuropathy ≥grade 2 according to NCI version 4.0 criteria.
* More than one previous line of chemotherapy in advanced setting.
* Concomitant hormonal therapy for MBC.
* Ongoing anti-coagulation therapy.
* Subjects of reproductive potential who are pregnant, breast feeding or not willing to use effective contraceptive precautions during the study and for at least one month after the last dose of investigational product in the judgment of the investigator.
* Patients with psychiatric disorder or other disease leading to incompliance to the therapy.
* Known hypersensitivity to any ingredient of the study drug.
* An interval of less than 3 weeks between the last dose of previous chemotherapy and randomization.
* Previous treated by oral NVB.
* Treatment with any investigational drug within 30 days before the beginning of treatment with study drug. Less than 30 days since receipt of any other investigational product or device.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2019-02-20 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | 12 weeks
  Disease Control Rate (DCR) is the proportion of subjects who have best overall response of CR + PR + SD with duration of ≥6 weeks.

SECONDARY OUTCOMES:
Time to Tumor Progression | up to 36 months
  Time to Tumor Progression (TTP) is defined as the time from randomization to time of progressive disease.
Time to Treatment Failure | up to 36 months
  Time to Treatment Failure (TTF) is defined as the time from randomization to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient toxicity, patient preference, or death.
Progression free survival | up to 36 months
  Progression free survival (PFS) is the time from the date of randomization to the date of first documentation of disease progression, or to the date of death from any case, whichever occurs first.
Overall survival | up to 60 months
  Overall survival (OS) will be measured from the date of randomization until the date of death from any case.
Adverse events | up to 36 months
  Adverse events including Serious AEs and non-serious AEs (since ICF signed and until 30 days after last intake of study medication)
Quality of Life (QoL) | up to 36 months
  The FACT-B +4 (Version 4) (Appendix ) QoL questionnaires will be filled in at baseline before randomization, then every 6 weeks during the Randomization Treatment Period and at EoTV. Changes of the scores from baseline of the parameters will be provided from baseline.